CLINICAL TRIAL: NCT05261555
Title: Acceptability and Usability of a Mobile Health App for Family Obesity Prevention and Management: A Mixed-methods Feasibility Study
Brief Title: Mixed Methods Feasibility Study of an App for Childhood Obesity Prevention and Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Collaborators: Health Education England, Wessex (Other)
Responsible Party: Principal Investigator, Edward Meinert, PhD, Associate Professor of eHealth, University of Plymouth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R62092/RE001
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Child Obesity
Keywords: child obesity; digital health; mobile applications; behavior change
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Using the NoObesity app (Experimental): A mobile digital app ("NoObesity") that enables families to set goals, track progress, play games, and access additional information and healthcare professionals to access training and monitor patients' progress.
  Interventions: Device: NoObesity app

INTERVENTIONS:
Device: NoObesity app — The NoObesity system consists of two linked apps - the NoObesity Family app and the NoObesity Professional app.

SUMMARY:
This evaluation evaluated Health Education England's NoObesity digital health app's usability and acceptability to undertake activities improving families' diet, physical activity and weight. The purpose of the study is to evaluate the app's influence on self-efficacy and goal setting and to determine what can be learned to improve its design for future studies, should there be evidence of adoption and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* adult users (over 18 years)
* fluent in English
* willing to use the app
* parents or legal guardians of a child or children OR health care professionals linked to the parent or guardian
* owner of a smartphone to access the app, with 4G data access

Exclusion Criteria:

* individuals who are known to the researchers or staff at Health Education England
* deaf or hearing impairment
* prior use of the app before study commencement
* refusal to give informed consent
* children, vulnerable young people, or vulnerable adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2020-06-27 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
User experiences and acceptability of the NoObesity app | 6 months
  Measured qualitatively through semi-structured interviews to examine what participants liked, disliked, and what they thought could be improved

SECONDARY OUTCOMES:
Usability of the NoObesity app | 6 months
  Measured using the System Usability Scale (minimum of 0, maximum of 100, higher scores indicate better usability)
Qualitative user perspectives of usability | 6 months
  Qualitative feedback from semi-structured interviews
Perceived impact of app on motivation | 6 months
  Qualitative feedback from semi-structured interviews
Perceived impact of specific app features on motivation | 6 months
  Measured quantitatively on self-report final survey
Perceived impact of app on health behaviours | 6 months
  Qualitative feedback from semi-structured interviews
Self-reported impact of the app on health behaviours | 6 months
  Measured quantitatively on self-report final survey
Perceived impact of app on self-efficacy | 6 months
  Measured quantitatively by assessing users' confidence in their ability to achieve goals in the app and in the final survey
Engagement with the app | 6 months
  Measured using app use data (first and last logins) and self-reported engagement with the app
Factors relating to adoption, implementation, and sustainability | 6 months
  Measured qualitatively in semi-structured interviews with participants and representatives from Health Education England

CONTACTS AND LOCATIONS:
Overall Officials: Edward Meinert, PhD, Principal Investigator — University of Plymouth
Locations (1):
- University of Plymouth, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meinert E, Rahman E, Potter A, Lawrence W, Van Velthoven M. Acceptability and Usability of the Mobile Digital Health App NoObesity for Families and Health Care Professionals: Protocol for a Feasibility Study. JMIR Res Protoc. 2020 Jul 22;9(7):e18068. doi: 10.2196/18068. PMID 32706703
- [Derived] Milne-Ives M, Homer SR, Andrade J, Meinert E. Mapping the Process of Engagement With Digital Health Interventions: A Cross-Case Synthesis. Mayo Clin Proc Innov Qual Outcomes. 2025 May 27;9(3):100625. doi: 10.1016/j.mayocpiqo.2025.100625. eCollection 2025 Jun. PMID 40503087
- [Derived] Milne-Ives M, Rahman E, Bradwell H, Baines R, Boey T, Potter A, Lawrence W, Helena van Velthoven M, Meinert E. Barriers and facilitators to parents' engagement with and perceived impact of a childhood obesity app: A mixed-methods study. PLOS Digit Health. 2024 Mar 27;3(3):e0000481. doi: 10.1371/journal.pdig.0000481. eCollection 2024 Mar. PMID 38536852